CLINICAL TRIAL: NCT02173548
Title: Interleukin-1 Blockade in Heart Failure With Preserved Ejection Fraction (HFpEF): a Randomized Placebo-controlled Double Blinded Study (D-HART2)
Brief Title: Interleukin-1 Blockade in HF With Preserved EF
Acronym: D-HART2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20000118; 1R34HL118348-01A1 (NIH)
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: heart failure; HFpEF; diastole; diastolic heart failure; inflammation; interleukin-1; C-reactive protein
MeSH Terms: conditions — Heart Failure; Heart Murmurs; Heart Failure, Diastolic; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anakinra (Active Comparator): Anakinra 100 mg given subcutaneously once daily for 12 weeks
  Interventions: Drug: Anakinra
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra
  Other Names: Kineret
  Arms: Anakinra
Drug: Placebo
  Arms: Placebo

SUMMARY:
* Heart Failure with Preserved Ejection Fraction (HFpEF) is a common form of heart failure
* Standard treatment for heart failure, show less than ideal results in HFpEF
* Evidence of systemic inflammation is common in all forms of heart failure, including HFpEF
* The main hypothesis of this study is that systemic inflammation contributes to heart failure symptoms and exercise limitations in patients with HFpEF
* The main objective is to treat patients with HFpEF and evidence of systemic inflammation with an anti-inflammatory drug targeting Interleukin-1 (or placebo) to determine effects on cardiovascular function

DETAILED DESCRIPTION:
Heart Failure with Preserved Ejection Fraction (HFpEF) is a common form of heart failure, characterized by symptoms of congestion and impaired exercise tolerance, secondary to impaired left ventricular filling (diastole) in absence of a significant impairment in contractility (LVEF>50%) or significant valvular abnormalities, shunts or intra- or extra-cavitary obstruction.

The standard treatment for patient with heart failure is very effective in Heart Failure with Reduced Ejection Fraction (HFrEF), but it not very effective in HFpEF.

Evidence of systemic inflammation is common in all forms of heart failure, including HFpEF, and predicts worse outcomes. C reactive protein (CRP) is the preferred inflammatory biomarker used as risk predictor for cardiovascular disease. Patients with heart failure (HFpEF or HFrEF) with elevated CRP levels are more likely to be severely limited by heart failure symptoms, are more likely to be admitted to the hospital for heart failure, and are more likely to die of cardiac causes.

Preclinical studies show that a key mediator of systemic inflammation, Interleukin-1 (IL-1), impairs cardiac and vascular function, and may contribute to the pathogenesis of heart failure.

The main hypothesis of this study is that systemic inflammation, and IL-1 in particular, contributes to heart failure symptoms and exercise limitations in patients with HFpEF.

The main objective is to treat patients with HFpEF and evidence of systemic inflammation with an IL-1 blocker, anakinra (recombinant human IL-1 receptor antagonist)(or placebo) to determine effects on exercise capacity measured as peak oxygen consumption at maximal cardiopulmonary exercise testing.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms and signs of heart failure (NYHA II-III) and prior hospitalization for heart failure
2. Recent Imaging Study (<12 months) showing LVEF>50% and Left Ventricular End Diastolic Volume Index (LVEDVI) <97ml/m2
3. Evidence of abnormal LV relaxation, filling, diastolic distensibility, and diastolic stiffness as shown by one of the following

   a. Invasive Hemodynamic measurements i. mean Pulmonary Capillary Wedge Pressure (mPCW) >12 ii. Left Ventricular End Diastolic Pressure (LVEDP) >16 mmHg b. Tissue Doppler Echocardiogram i. E/E' >15 ii. E/E' 8-15 and one of the following: Left Ventricular Hypertrophy (LVH), Atrial fibrillation, Left Atrial Enlargement (LAE), E/A <0.5 + DT (Deceleration Time) >280, c. Biomarkers i. Brain Natriuretic Peptide (BNP) >200pg/ml (not due to a concomitant disease such as pulmonary arterial hypertension, pulmonary embolism, acute renal failure, or other)
4. CRP > 2.0 mg/L

Exclusion Criteria:

* Age <21
* Concomitant conditions or treatments which would affect completion of the study or interpretation of the study tests including but not limited to the following conditions:

  * physical inability to walk or run on a treadmill
  * angina or evidence of spontaneous or inducible ischemia
  * uncontrolled arterial hypertension
  * atrial fibrillation (or other arrhythmias)
  * moderate to severe valvular heart disease
  * chronic pulmonary disease
  * anemia (Hgb<10 g/dl)
* Angina, uncontrolled hypertension or electrocardiograph (ECG) changes (i.e. ischemia, arrhythmias) that limit maximum exertion during cardiopulmonary exercise testing
* Anticipated need for cardiac resynchronization therapy (CRT) or automated-implantable cardioverter defibrillator (AICD) or coronary revascularization or cardiac surgery
* Active infection including chronic infection
* Active cancer (or prior diagnosis of cancer within the past 10 years)
* Recent (<14 days) or active use of immunosuppressive drugs (including but not limited to high-dose corticosteroids [>1_mg/kg of prednisone equivalent], Tumor Necrosis Factor (TNF)-α blockers, cyclosporine) not including Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) or corticosteroids used for IV dye allergy only)
* Chronic auto-immune or auto-inflammatory disease (including but not limited to rheumatoid arthritis, systemic lupus erythematosus)
* Neutropenia (absolute neutrophil count<1,800/mm3 [or <1,000/mm3 in African-American patients])
* Severe impairment in renal function (estimated glomerular filtration rate <30 ml/kg*min)
* Recent or planned use of vaccination with live attenuated viruses
* Allergy to rubber or latex
* Allergy to products derived from Escherichia coli
* Pregnancy or breastfeeding
* Inability to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04-11 (Actual); Study Completion 2017-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University; Benjamin Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Van Tassell BW, Trankle CR, Canada JM, Carbone S, Buckley L, Kadariya D, Del Buono MG, Billingsley H, Wohlford G, Viscusi M, Oddi-Erdle C, Abouzaki NA, Dixon D, Biondi-Zoccai G, Arena R, Abbate A. IL-1 Blockade in Patients With Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2018 Aug;11(8):e005036. doi: 10.1161/CIRCHEARTFAILURE.118.005036. PMID 30354558
- [Derived] Van Tassell BW, Buckley LF, Carbone S, Trankle CR, Canada JM, Dixon DL, Abouzaki N, Oddi-Erdle C, Biondi-Zoccai G, Arena R, Abbate A. Interleukin-1 blockade in heart failure with preserved ejection fraction: rationale and design of the Diastolic Heart Failure Anakinra Response Trial 2 (D-HART2). Clin Cardiol. 2017 Sep;40(9):626-632. doi: 10.1002/clc.22719. Epub 2017 May 5. PMID 28475816

RESULTS

PARTICIPANT FLOW:
Groups:
- Anakinra: Anakinra 100 mg given subcutaneously once daily for 12 weeks
  Anakinra
- Placebo: Matching Placebo
  Placebo
Period: Overall Study
Arm/Group | Anakinra | Placebo
Started | 21 | 10
Completed | 20 | 8
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra | Placebo | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 10 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 5 | 18
  Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Aerobic Exercise Capacity
Description: Absolute changes in aerobic exercise capacity (peak VO2) after 12 weeks treatment. This will compare patients treated with anakinra and provide a randomized, double-blinded assessment of the effects of IL-1β blockade on aerobic exercise performance.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: ml/kg/min
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 20 | 8
ml/kg/min | -0.2 [-0.9 to 1.7] | 1.0 [-1.3 to 2.0]

2. Primary Outcome: Change in Ventilatory Eefficiency
Description: Absolute changes in ventilatory efficiency (VE/VCO2 [carbon dioxide] slope) after 12 weeks treatment. This will compare patients treated with anakinra vs placebo, and provide a randomized, double-blinded assessment of the effects of IL-1β blockade on aerobic exercise performance.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: VE/VO2 slope
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 20 | 8
VE/VO2 slope | 0.2 [-2.1 to 1.8] | -0.2 [-1.6 to 1.3]

3. Secondary Outcome: Echocardiographic Assessment of Diastolic and Systolic Function (Left Ventricular Ejection Fraction)
Description: Structural and functional echocardiographic parameters include left and right ventricular dimensions, mass, systolic and diastolic function. (Change in e')
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: cm/second
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 20 | 8
cm/second | 0.3 [-0.8 to 1.0] | 1.9 [-0.3 to 4.0]

4. Secondary Outcome: Change in Diastolic and Contractile Reserve (e' Velocity and E/e' Ratio)
Description: Exercise stress echocardiography will be performed at baseline and 12 weeks to measure diastolic and contractile reserve. We will perform an assessment before initiation of exercise and immediately after cessation of peak exercise.
Time Frame: Baseline to 12 weeks
Population: Data not available for all participants.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 8 | 3
ratio | -0.7 [-5.7 to 3.1] | 0.7 [-4.5 to 0.7]

5. Secondary Outcome: Change in Inflammation (C Reactive Protein Levels)
Description: The change C reactive protein (CRP) levels will be reported at 12 weeks. Higher C reactive protein levels indicate greater inflammation.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: mg/l
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 20 | 8
mg/l | -2.8 [-7.5 to -0.5] | 1.2 [-1.2 to 2.4]

6. Secondary Outcome: Change in Quality of Life Questionnaire-Minnesota Living With Heart Failure Questionnaire (MLWHF)
Description: The Minnesota Living with Heart Failure questionnaire (MLWHF) is a 21-question graded questionnaire that has been extensively used to measure impairment in quality of life in patients with HF, with higher scores reflecting increased burden of HF symptoms. The questionnaire will be administered in accordance with cardiopulmonary test (CPET) and echocardiography. Scores range from zero to 105 with lower scores indicating better quality of life.
Time Frame: Baseline to 24 weeks
Measure: Median (Inter-Quartile Range); unit: units on MWLHF scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 20 | 8
units on MWLHF scale | -6 [-19 to 1] | -16 [-24 to -11]

7. Secondary Outcome: Change in Quality of Life Questionnaire-Duke Activity Status Index (DASI)
Description: Two independent questionnaires will be used to assess quality of life and HF symptoms. The Duke Activity Status Index (DASI) questionnaire is a 12-question, yes/no, instrument that allows for the calculation of perceived functional capacity, in which each question describes a different physical activity and the questions are weighted according to their degree of physical exertion. Higher scores indicate greater functional capacity. The questionnaire will be administered at 0, 4, 12 and 24 weeks in accordance with cardiopulmonary test (CPET) and echocardiography. Scores range from zero to 58.2 with higher scores indicating higher functional status.
Time Frame: Baseline to 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on DASI scale
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 20 | 8
units on DASI scale | 4 [-2.5 to 12.6] | 6.5 [-6.6 to 11.4]

8. Secondary Outcome: Hospital Admission for Acute Decompensated Heart Failure
Description: Number of participants admitted to hospital for acute decompensated heart failure
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 20 | 8
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: One participant in the anakinra arm withdrew from the study before receiving any study-related interventions.
Arm/Group | Anakinra | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/10
Other Adverse Events (participants affected / at risk) | 4/20 | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=20) | Placebo (N=10)
Acute decompensated heart failure (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=20) | Placebo (N=10)
Upper respiratory infection (Infections and infestations) | 1 (1) | 2 (2)
Non serious infection (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT02173548/Prot_SAP_000.pdf